CLINICAL TRIAL: NCT03953586
Title: Hysteroscopic Bubble Suction Test and Tubal Peristalsis (Darwish Test) in Hydrosalpnix
Status: Completed | Type: Observational
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Professor Atef Darwish, Professor of Obstetrics and Gynecology, Assiut University, Assiut, Egypt, Woman's Health University Hospital, Egypt
Other Study IDs: WomansHealthUHEgypt
Record Dates: First submitted 2019-05-12; First posted 2019-05-16 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Tubal Patency
Keywords: laparoscopy; hysteroscopy,; tubal patency,; bubble test,; peristalsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bubble suction test and peristalsis in hydrosalpnix: . Group A: Women with unilateral or bilateral blockage of the distal end of the fallopian tubes with tubal distension.
  Interventions: Diagnostic Test: Bubble suction test and tubal peristalsis
- bubble suction test and peristalsis in normal tubes: Group B: Women with normal appearance of the fallopian tubes by HSG.
  Interventions: Diagnostic Test: Bubble suction test and tubal peristalsis

INTERVENTIONS:
Diagnostic Test: Bubble suction test and tubal peristalsis — Efficacy of this test in cases of hydrosalpnix (group A) and normal tubes (group B)

SUMMARY:
Tubal patency testing is essential for infertility evaluation. Standard tests are hysterosalpingography and laparoscopic perchromation test. In 2016, a hysteroscopic bubble suction test was described in apparently normal tubes. However, the efficacy of bubble suction test in abnormal tubes like hydrosalpnix has not been studied.

DETAILED DESCRIPTION:
Nowadays, hysteroscopy is extensively used for fertility assessment. In a previous study, it is recommended to add hysteroscopy to the routine infertility work-up to achieve a better assessment of infertility cases.

In 2016, hysteroscopy as a predictor test of tubal patency and tubal peristalsis was introduced. It is concluded that hysteroscopic bubble suction test is a good initial screening test for tubal patency nearly comparable to HSG and DL. It should be attempted in every case of OH prior to referral for more invasive HSG or laparoscopic chromopertubation test.

Thereafter, some authors tried the same idea of bubble suction test and were over-enthusiastic with this test and considered it superior to hysterosalpingography (HSG) in detection of tubal patency in infertile women. They wrongly described HSG as a historic tool despite being recommended as a basic infertility test by many organizations. Some authors criticized the results of these studies and underestimated their clinical implication. One of the objections were lack of differentiation between normal tubes and damaged or narrowed but still patent tubes.

Aim of the work:

To test whether bubble suction test and osteal peristalsis are preserved or lost in cases with hydrosalpnix.

Design: A prospective double blinded randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Infertility patients scheduled for combined laparoscopy and hysteroscopy

Exclusion Criteria:

* No HSG

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women with a history of HSG
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
percentage of positive tests in both pathologic and healthy tubes | 6 months
  Bubble suction test+ tubal peristalsis

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes